CLINICAL TRIAL: NCT04269200
Title: A Randomised, Multicentre, Double-blind, Placebo-controlled, Phase III Study of First-line Carboplatin and Paclitaxel in Combination With Durvalumab, Followed by Maintenance Durvalumab With or Without Olaparib in Patients With Newly Diagnosed Advanced or Recurrent Endometrial Cancer (DUO-E)
Brief Title: Durvalumab With or Without Olaparib as Maintenance Therapy After First-Line Treatment of Advanced and Recurrent Endometrial Cancer
Acronym: DUO-E
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: The Gynecologic Oncology Group (GOG) Foundation Inc (Unknown); The European Network for Gynaecological Oncological Trial groups (ENGOT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9311C00001; GOG-3041 (Other: Gynecologic Oncology Group(GOG) Foundation Inc); ENGOT-EN10 (Other: The European Network for Gynaecological Oncological Trial groups); D9311C00001 (Other: AZ DCode); 2022-502746-27-00 (Registry Identifier: CTIS (EU)); 2019-004112-60 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Neoplasms
Keywords: Cancer of Endometrium; Cancer of the Endometrium; Carcinoma of Endometrium; Endometrial Cancer; Endometrial Carcinoma; Endometrium Cancer; Neoplasms, Endometrial
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib; durvalumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (control) (Active Comparator): Platinum-based chemotherapy and durvalumab placebo followed by maintenance durvalumab placebo and olaparib placebo (tablets).
  Interventions: Drug: durvalumab placebo; Drug: olaparib placebo; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (durvalumab+placebo) (Experimental): Platinum-based chemotherapy and durvalumab followed by maintenance durvalumab and olaparib placebo
  Interventions: Biological: durvalumab; Drug: olaparib placebo; Drug: Carboplatin; Drug: Paclitaxel
- Arm C (durvalumab+olaparib) (Experimental): Platinum-based chemotherapy and durvalumab followed by maintenance durvalumab and olaparib.
  Interventions: Drug: olaparib; Biological: durvalumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: olaparib — Olaparib tablets
  Arms: Arm C (durvalumab+olaparib)
Biological: durvalumab — Durvalumab by intravenous infusion
  Arms: Arm B (durvalumab+placebo); Arm C (durvalumab+olaparib)
Drug: durvalumab placebo — Matching placebo for intravenous infusion
  Arms: Arm A (control)
Drug: olaparib placebo — Placebo tablets to match olaparib
  Arms: Arm A (control); Arm B (durvalumab+placebo)
Drug: Carboplatin — Standard of care chemotherapy
Drug: Paclitaxel — Standard of care chemotherapy

SUMMARY:
A study to assess the efficacy and safety of durvalumab in combination with platinum-based chemotherapy (paclitaxel + carboplatin) followed by maintenance durvalumab with or without olaparib for patients with newly diagnosed advanced or recurrent endometrial cancer.

DETAILED DESCRIPTION:
This Phase III study will assess the efficacy and safety of durvalumab in combination with platinum-based chemotherapy (paclitaxel + carboplatin) followed by maintenance durvalumab with or without olaparib for patients with newly diagnosed advanced or recurrent endometrial cancer.

Target patient population: Adult female patients with histologically confirmed diagnosis of epithelial endometrial carcinoma (excluding sarcomas): newly diagnosed Stage III, newly diagnosed Stage IV, or recurrent endometrial cancer

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of screening and female.
* Histologically confirmed diagnosis of epithelial endometrial carcinoma. All histologies, including carcinosarcomas, will be allowed. Sarcomas will not be allowed.
* Patient must have endometrial cancer in one of the following categories:

  1. Newly diagnosed Stage III disease (measurable disease per RECIST 1.1 following surgery or diagnostic biopsy),
  2. Newly diagnosed Stage IV disease (with or without disease following surgery or diagnostic biopsy)
  3. Recurrence of disease (measurable or non-measurable disease per RECIST 1.1) where the potential for cure by surgery alone or in combination is poor.
* Naïve to first line systemic anti-cancer treatment. For patients with recurrent disease only, prior systemic anti-cancer treatment is allowed only if it was administered in the adjuvant setting and there is at least 12 months from date of last dose of systemic anti-cancer treatment administered to date of subsequent relapse
* FPPE tumor sample must be available for MMR evaluation.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days of starting study treatment.

Exclusion Criteria:

* History of leptomeningeal carcinomatosis.
* Brain metastases or spinal cord compression.
* Prior treatment with PARP inhibitors.
* Any prior exposure to immune-mediated therapy, including (but not limited to) other anti CTLA-4, anti-PD-1, anti-PD-L1, or anti-programmed-cell-death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.

Ages: 18 Years to 150 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects only
Enrollment: 805 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2027-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N. Westin, MD, MPH, FACOG, Principal Investigator — M.D. Anderson Cancer Center
Locations (168):
- United States (48):
  - Research Site, Tucson, Arizona
  - Research Site, Concord, California
  - Research Site, La Jolla, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Aurora, Colorado
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Tampa, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Arlington Heights, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Saint Paul, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Lebanon, New Hampshire
  - Research Site, Camden, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, New York, New York
  - Research Site, Pinehurst, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Tigard, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tyler, Texas
  - Research Site, Webster, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Australia (5):
  - Research Site, Clayton
  - Research Site, Malvern
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Sydney
- Belgium (9):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Libramont-Chevigny
  - Research Site, Liège
- Brazil (8):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Passo Fundo
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (19):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangdong
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Pereira
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (5):
  - Research Site, Bonn
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Leipzig
- Greece (3):
  - Research Site, Athens
  - Research Site, Chaïdári
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Szolnok
- India (2):
  - Research Site, Hisar
  - Research Site, Mumbai
- Israel (5):
  - Research Site, Be’er Ya‘aqov
  - Research Site, Hadera
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Tel Aviv
- Japan (17):
  - Research Site, Chūōku
  - Research Site, Kashiwa-shi
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Nakagami-gun
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Toon-Shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Oaxaca City
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
- Russia (7):
  - Research Site, Anzorey
  - Research Site, Kazan, Tatarstan
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saransk
  - Research Site, Sochi
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Yangsan
- Spain (6):
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Girona
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Mallorca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Nishio S, Nishikawa T, Mori M, Kamiura S, Sumi T, Yunokawa M, Imai Y, Kondo E, Takehara K, Takano H, Kudaka W, Kado N, Yamagami W, Kato H, Nishino K, Usami T, Hamanishi J, Nii M, Takaya I, Okamoto A. Durvalumab plus carboplatin/paclitaxel followed by durvalumab with or without olaparib as first-line treatment for newly diagnosed advanced or recurrent endometrial cancer: Japan subset from the phase III DUO-E trial. J Gynecol Oncol. 2025 Jul;36(4):e118. doi: 10.3802/jgo.2025.36.e118. PMID 40590327
- [Derived] Bogani G, Monk BJ, Powell MA, Westin SN, Slomovitz B, Moore KN, Eskander RN, Raspagliesi F, Barretina-Ginesta MP, Colombo N, Mirza MR. Adding immunotherapy to first-line treatment of advanced and metastatic endometrial cancer. Ann Oncol. 2024 May;35(5):414-428. doi: 10.1016/j.annonc.2024.02.006. Epub 2024 Feb 29. PMID 38431043
- [Derived] Westin SN, Moore K, Chon HS, Lee JY, Thomes Pepin J, Sundborg M, Shai A, de la Garza J, Nishio S, Gold MA, Wang K, McIntyre K, Tillmanns TD, Blank SV, Liu JH, McCollum M, Contreras Mejia F, Nishikawa T, Pennington K, Novak Z, De Melo AC, Sehouli J, Klasa-Mazurkiewicz D, Papadimitriou C, Gil-Martin M, Brasiuniene B, Donnelly C, Del Rosario PM, Liu X, Van Nieuwenhuysen E; DUO-E Investigators. Durvalumab Plus Carboplatin/Paclitaxel Followed by Maintenance Durvalumab With or Without Olaparib as First-Line Treatment for Advanced Endometrial Cancer: The Phase III DUO-E Trial. J Clin Oncol. 2024 Jan 20;42(3):283-299. doi: 10.1200/JCO.23.02132. Epub 2023 Oct 21. PMID 37864337
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9311C00001&attachmentIdentifier=911f5098-85b6-4bc7-a5ed-a96253cccca6&fileName=D9311C00001_16.1.9_Statistical_Methods_and_Analysis-final-4.0_for_RRF.pdf&versionIdentifier=
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9311C00001&attachmentIdentifier=aadf8b74-3143-4698-87a8-919885a5487a&fileName=d9311c00001-csp-v6_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9311C00001&attachmentIdentifier=40f19bd2-bcd3-443f-8eab-09293f2ec2fb&fileName=d9311c00001-study-synopsis-china_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9311C00001&attachmentIdentifier=0b345ab2-2cb9-45b1-8127-5e84e448ac9a&fileName=d9311c00001-study-synopsis-global_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global Cohort: 875 patients screened across 179 centres in 22 countries; 718 were randomised. Results were reported for analysis of progression-free survival (PFS) (data cut-off [DCO]: 12 Apr 2023).
  China Cohort: 172 patients screened across 25 sites; 129 were randomized. Results were reported for analysis of PFS (DCO: 08 Jul 2024).
  In total, 805 patients were randomised; 718 to the Global cohort, 129 to the China cohort, with 42 patients overlapping and belonging to both cohorts.
Pre-assignment Details: It was planned that approximately 699 women from the Global cohort and 129 women from the China cohort, with newly diagnosed advanced or recurrent endometrial cancer, were to receive durvalumab/placebo in combination with platinum-based chemotherapy followed by maintenance durvalumab/placebo (same treatment as during chemotherapy phase) and olaparib/placebo in a 1:1:1 ratio.
Groups:
- Standard of Care (SoC): Platinum-based chemotherapy (paclitaxel and carboplatin) every 3 weeks (Q3W) for a maximum of 6 cycles with durvalumab placebo (intravenous [IV]) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received durvalumab placebo (IV) every 4 weeks (Q4W) and olaparib placebo (tablets) twice daily (bd) orally as maintenance treatment until disease progression.
- SoC + Durvalumab: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
- SoC + Durvalumab + Olaparib: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with 300 mg olaparib (tablets) bd orally as maintenance treatment until disease progression.
Period: Global Cohort
Arm/Group | Standard of Care (SoC) | SoC + Durvalumab | SoC + Durvalumab + Olaparib
Started | 241 | 238 | 239
Completed (Patients ongoing study at time of primary PFS analysis DCO: 12 Apr 2023) | 147 | 159 | 170
Not Completed | 94 | 79 | 69
Not completed — Death | 72 | 54 | 49
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 22 | 25 | 18
Period: China Cohort
Arm/Group | Standard of Care (SoC) | SoC + Durvalumab | SoC + Durvalumab + Olaparib
Started | 44 | 43 | 42
Completed (Patients ongoing study at time of primary PFS analysis DCO: 08 Jul 2024) | 30 | 29 | 24
Not Completed | 14 | 14 | 18
Not completed — Death | 12 | 11 | 13
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Global cohort: 241 SoC, 238 SoC + Durvalumab, 239 SoC + Durvalumab + Olaparib China cohort: 44 SoC, 43 SoC + Durvalumab, 42 SoC + Durvalumab + Olaparib
  There were 42 patients included in both Global and China cohorts (15 SOC, 14 SoC + Durvalumab, 13 SoC + Durvalumab + Olaparib).
Groups:
- SoC (Global Cohort & China Cohort): Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with durvalumab placebo (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received durvalumab placebo (IV) Q4W and olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
- SoC + Durvalumab (Global Cohort & China Cohort): Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
- SoC + Durvalumab + Olaparib (Global Cohort & China Cohort): Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with 300 mg olaparib (tablets) bd orally as maintenance treatment until disease progression.
- Total: Total of all reporting groups
Arm/Group | SoC (Global Cohort & China Cohort) | SoC + Durvalumab (Global Cohort & China Cohort) | SoC + Durvalumab + Olaparib (Global Cohort & China Cohort) | Total
Number analyzed (Participants) | 270 | 267 | 268 | 805
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening Population: The results are presented by Global cohort and by China cohort.
  Years
    Global cohort: number analyzed (Participants) | 241 | 238 | 239 | 718
    Global cohort | 62.1 (10.36) | 63.3 (9.82) | 62.4 (9.90) | 62.6 (10.03)
    China cohort: number analyzed (Participants) | 44 | 43 | 42 | 129
    China cohort | 58.3 (8.73) | 57.6 (10.57) | 59.3 (8.41) | 58.4 (9.24)
Age, Customized [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort.
  Participants
    Global cohort: number analyzed (Participants) | 241 | 238 | 239 | 718
    Global cohort: <65 years | 124 | 122 | 135 | 381
    Global cohort: >=65 years | 117 | 116 | 104 | 337
    China cohort: number analyzed (Participants) | 44 | 43 | 42 | 129
    China cohort: <65 years | 35 | 30 | 30 | 95
    China cohort: >=65 years | 9 | 13 | 12 | 34
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort.
  Participants
    Global cohort: number analyzed (Participants) | 241 | 238 | 239 | 718
    Global cohort: Female | 241 | 238 | 239 | 718
    China cohort: number analyzed (Participants) | 44 | 43 | 42 | 129
    China cohort: Female | 44 | 43 | 42 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort.
  Participants
    Global cohort: number analyzed (Participants) | 241 | 238 | 239 | 718
    Global cohort: Hispanic or Latino | 20 | 28 | 32 | 80
    Global cohort: Not Hispanic or Latino | 218 | 208 | 206 | 632
    Global cohort: Unknown or Not Reported | 3 | 2 | 1 | 6
    China cohort: number analyzed (Participants) | 44 | 43 | 42 | 129
    China cohort: Hispanic or Latino | 0 | 0 | 0 | 0
    China cohort: Not Hispanic or Latino | 44 | 43 | 42 | 129
    China cohort: Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort.
  Participants
    Global cohort: number analyzed (Participants) | 241 | 238 | 239 | 718
    Global cohort: White | 143 | 136 | 133 | 412
    Global cohort: Asian | 73 | 72 | 70 | 215
    Global cohort: Black or African American | 10 | 11 | 14 | 35
    Global cohort: Other | 10 | 8 | 12 | 30
    Global cohort: American Indian or Alaska Native | 0 | 6 | 6 | 12
    Global cohort: Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
    Global cohort: Not reported | 3 | 5 | 3 | 11
    China cohort: number analyzed (Participants) | 44 | 43 | 42 | 129
    China cohort: White | 0 | 0 | 0 | 0
    China cohort: Asian | 44 | 43 | 42 | 129
    China cohort: Black or African American | 0 | 0 | 0 | 0
    China cohort: Other | 0 | 0 | 0 | 0
    China cohort: American Indian or Alaska Native | 0 | 0 | 0 | 0
    China cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    China cohort: Not reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to RECIST 1.1, Based on Investigator Assessments
Description: To demonstrate the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy by assessment of PFS (using investigator assessment according to Response Evaluation Criteria in Solid Tumours version 1.1 [RECIST 1.1]) in patients with newly diagnosed advanced or recurrent endometrial cancer
Time Frame: At baseline, every 9 weeks (wks) up to 18 wks, then every 12 wks until objective radiological disease progression. Assessed until 12 Apr 2023 DCO (08 Jul 2024 DCO for China cohort), up to 50 months
Population: Full Analysis Set (FAS) consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). China FAS includes all patients who were randomised at sites in China and Hong Kong.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Cohort - SoC; China Cohort - SoC: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with durvalumab placebo (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received durvalumab placebo (IV) Q4W and olaparib placebo (tablets) twice bd orally as maintenance treatment until disease progression.
- Global Cohort - SoC + Durvalumab; China Cohort - SoC + Durvalumab: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
- Global Cohort - SoC + Durvalumab + Olaparib; China Cohort - SoC + Durvalumab + Olaparib: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, patients without objective disease progression received 1500 mg durvalumab (IV) Q4W with 300 mg olaparib (tablets) bd orally as maintenance treatment until disease progression.
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 241 | 238 | 239 | 44 | 43 | 42
Months | 9.6 [9.0 to 9.9] | 10.2 [9.7 to 14.7] | 15.1 [12.6 to 20.7] | 9.7 [7.6 to 12.3] | 9.9 [8.2 to 20.6] | 9.9 [7.1 to 12.6]
Statistical Analysis 1: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab; Test type: Superiority; p = 0.003, Regression, Cox — Determined using a log-rank test stratified by mismatch repair (MMR) status (proficient versus deficient) and disease status (recurrent versus newly diagnosed); Model was stratified by MMR status (proficient versus deficient) and disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.57 to 0.89] — A hazard ratio less than 1 favours SoC + Durvalumab
Statistical Analysis 2: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by MMR status (proficient versus deficient) and disease status (recurrent versus newly diagnosed); Model was stratified by MMR status (proficient versus deficient) and disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.43 to 0.69] — A hazard ratio less than 1 favours SoC + Durvalumab + Olaparib
Statistical Analysis 3: Comparison: China Cohort - SoC vs China Cohort - SoC + Durvalumab; Test type: Superiority; Regression, Cox — China cohort designed to provide descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.42 to 1.25] — A hazard ratio less than 1 favours SoC + Durvalumab
Statistical Analysis 4: Comparison: China Cohort - SoC vs China Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Regression, Cox — China cohort designed to provide descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.57 to 1.61] — A hazard ratio less than 1 favours SoC + Durvalumab + Olaparib

2. Secondary Outcome: Overall Survival (OS) Analysis
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of OS
Time Frame: Survival assessed every 2 months after RECIST defined radiological progression; assessed through study completion, up to 83 months
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Time From Randomisation to Second Progression or Death (PFS2) Based on Local Standard Clinical Practice
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of PFS2
Time Frame: At baseline, every 9 to 18 wks, then every 12 wks until objective radiological disease progression. Assessments then per local practice every 12 wks until second progression. Assessed until 12Apr2023 DCO (08Jul2024 DCO for China cohort), up to 50 months
Population: FAS consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). China FAS includes all patients who were randomised at sites in China and Hong Kong.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Cohort - SoC: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with durvalumab placebo (IV) Q3W.
  Following completion of chemotherapy treatment, participants without objective disease progression received durvalumab placebo (IV) Q4W and olaparib placebo (tablets) twice bd orally as maintenance treatment until disease progression.
- Global Cohort - SoC + Durvalumab: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, participants without objective disease progression received 1500 mg durvalumab (IV) Q4W with olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 241 | 238 | 239 | 44 | 43 | 42
Months | 19.1 [16.4 to 22.9] | 22.2 [18.7 to NA] — Insufficient PFS2 events to estimate upper confidence limit. | NA [NA to NA] — Insufficient PFS2 events to estimate median and confidence limits. | 24.2 [15.5 to NA] — Insufficient PFS2 events to estimate upper confidence limit. | 19.7 [15.3 to NA] — Insufficient PFS2 events to estimate upper confidence limit. | 15.3 [12.7 to NA] — Insufficient PFS2 events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab; Test type: Superiority; Regression, Cox — Descriptive analysis only; Model is unstratified; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.07] — A hazard ratio less than 1 favours SoC + Durvalumab
Statistical Analysis 2: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Regression, Cox — Descriptive analysis only; Model is unstratified; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.40 to 0.76] — A hazard ratio less than 1 favours SoC + Durvalumab + Olaparib
Statistical Analysis 3: Comparison: China Cohort - SoC vs China Cohort - SoC + Durvalumab; Test type: Superiority; Regression, Cox — China cohort designed to provide descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.48 to 2.21] — A hazard ratio less than 1 favours SoC + Durvalumab
Statistical Analysis 4: Comparison: China Cohort - SoC vs China Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Regression, Cox — China cohort designed to provide descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.68 to 2.90] — A hazard ratio less than 1 favours SoC + Durvalumab

4. Secondary Outcome: Objective Response Rate (ORR) Based on Investigator Assessment
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of ORR
Time Frame: At baseline, every 9 to 18 wks, then every 12 wks until objective radiological disease progression. Assessed until 12 Apr 2023 DCO (08 Jul 2024 DCO for China cohort), up to 50 months
Population: All participants with measurable disease at baseline were included in the analysis. FAS consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). China FAS includes all patients who were randomised at sites in China and Hong Kong. Odds ratio only calculated for Global cohort (per statistical analysis plan [SAP]).
Measure: Number; unit: Percentage of participants
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 198 | 202 | 184 | 37 | 32 | 33
Percentage of participants | 55.1 | 61.9 | 63.6 | 59.5 | 59.4 | 45.5
Statistical Analysis 1: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab; Test type: Superiority; Regression, Logistic — Descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.89 to 1.98] — An odds ratio greater than 1 favours SoC + durvalumab
Statistical Analysis 2: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Regression, Logistic — Descriptive analysis only; Model was stratified by disease status (recurrent versus newly diagnosed); Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.95 to 2.18] — An odds ratio greater than 1 favours SoC + durvalumab + Olaparib

5. Secondary Outcome: Duration of Response (DoR) Based on Investigator Assessment
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of DoR
Time Frame: At baseline, every 9 wks up to 18 wks, then every 12 wks until objective radiological disease progression. Assessed until 12 Apr 2023 DCO, up to 35 months
Population: All participants with confirmed response were included in the analysis. FAS consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). This endpoint was not assessed in the China cohort as it was not prespecified in the statistical analysis plan (SAP).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 109 | 125 | 117
Months | 7.7 [5.1 to 13.5] | 13.1 [6.0 to NA] — Insufficient DoR events to estimate upper confidence limit. | 21.3 [8.1 to 29.9]

6. Secondary Outcome: Time From Randomisation to First Subsequent Therapy or Death (TFST)
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of TFST
Time Frame: Time elapsed from randomisation to first subsequent therapy or death. Assessed every 12 wks following treatment discontinuation, through study completion (up to 83 months)
Reporting Status: Not Posted, anticipated posting 2027-06

7. Secondary Outcome: Time From Randomisation to Second Subsequent Therapy or Death (TSST)
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of TSST
Time Frame: Time elapsed from randomisation to second subsequent therapy or death. Assessed every 12 wks following treatment discontinuation, through study completion (up to 83 months)
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Time From Randomisation to Discontinuation of Treatment or Death (TDT)
Description: To determine the efficacy of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy in newly diagnosed advanced or recurrent endometrial cancer patients by assessment of TDT
Time Frame: Time elapsed from randomisation to study treatment discontinuation or death. Assessed through study completion, up to 83 months
Reporting Status: Not Posted, anticipated posting 2027-06

9. Secondary Outcome: Serum Concentration of Durvalumab
Description: To characterise the pharmacokinetics (PK) of durvalumab and durvalumab in combination with olaparib
Time Frame: PK sampling performed on Day 85 pre-dose, Day 183 pre-dose, and 3 months after study treatment discontinuation (up to 36 months)
Population: The Overall Number of Participants Analyzed reflects the total number of patients included in the PK Analysis Set, which comprises those treated with durvalumab per protocol and with valid PK data. However, PK concentrations were excluded at the sample level if they do not meet protocol-defined criteria. While some patients may not have any valid samples due to these exclusions, they remain part of the analysis population set by definition.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 204 | 213 | 36 | 35
μg/mL
  Day 85, pre-dose (Trough concentration): number analyzed (Participants) | 76 | 90 | 7 | 2
  Day 85, pre-dose (Trough concentration) | 203.133538 (32.6) | 196.218276 (31.7) | 183.414442 (32.7) | NA (NA) — As pre-specified in the Statistical Analysis Plan, three observations above the lower limit of quantification (LLOQ) are required as a minimum for a serum concentration to be summarised. Two observations above the LLOQ are presented as minimum and maximum with the other summary statistics as not calculated.
  Day 183, pre-dose (Trough concentration): number analyzed (Participants) | 26 | 35 | 0 | 1
  Day 183, pre-dose (Trough concentration) | 265.575840 (39.6) | 236.315365 (38.0) |  | NA (NA) — As pre-specified in the Statistical Analysis Plan, three observations above the lower limit of quantification (LLOQ) are required as a minimum for a serum concentration to be summarised. Two observations above the LLOQ are presented as minimum and maximum with the other summary statistics as not calculated.
  Follow-up 3-months (Last valid dose + 3 months): number analyzed (Participants) | 21 | 20 | 5 | 8
  Follow-up 3-months (Last valid dose + 3 months) | 27.977227 (104.4) | 14.031316 (206.8) | 33.310921 (43.0) | 11.252155 (1429.7)

10. Secondary Outcome: Anti-drug Antibodies (ADA) to Durvalumab
Description: To characterise the immunogenicity of durvalumab and durvalumab in combination with olaparib
Time Frame: Immunogenicity sampling performed on Day 1 pre-dose, Day 85 pre-dose, Day 183 pre-dose, and 3 and 6 months after study treatment discontinuation (up to 39 months)
Population: ADA Analysis Set. This includes all patients who receive at least 1 dose of durvalumab and have non-missing baseline ADA and at least 1 post-baseline ADA result.
Measure: Number; unit: Number of participants
Arm/Group | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 198 | 207 | 35 | 33
Number of participants
  ADA-positive at any visit (ADA prevalence) | 8 | 9 | 0 | 1
  Treatment-emergent ADA-positive (ADA incidence) | 2 | 0 | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0
  Treatment-induced ADA (positive post-baseline only) | 2 | 0 | 0 | 0
  ADA positive at baseline only | 6 | 9 | 0 | 1
  ADA positive post-baseline and positive at baseline | 0 | 0 | 0 | 0
  Persistently positive | 2 | 0 | 0 | 0
  Transiently positive | 0 | 0 | 0 | 0
  Neutralising antibody positive at any visit | 1 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Physical Functioning Score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients 30 (EORTC QLQ-C30)
Description: To determine effects on symptoms, functioning, and overall health related quality of life (HRQoL) of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy alone in newly diagnosed advanced or recurrent endometrial cancer patients. The physical functioning score is a score from 0 to 100. Higher scores on the physical functioning score indicate better health status/function.
Time Frame: At baseline, every 3 wks until Wk 18, and every 4 wks until the second progression. Assessed until 12 Apr 2023 DCO, up to 35 months. The average treatment effect over the first 12 months after randomisation is presented.
Population: FAS consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). All participants with a baseline and post baseline physical functioning score available were analysed. This endpoint was not assessed in the China cohort as it was not prespecified in the SAP.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 187 | 190 | 199
Score on a scale | -5.3 (1.03) | -3.6 (1.02) | -5.9 (0.98)
Statistical Analysis 1: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab; Test type: Superiority; Mixed model for repeated measures — Descriptive analysis only; Fixed effects for treatment, visit, and baseline score with the treatment by visit and baseline score by visit interaction. Random patient effect; Least-squares Mean Difference = 1.7, 95% CI 2-sided [-1.2 to 4.5]
Statistical Analysis 2: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Mixed model for repeated measures — Descriptive analysis only; [statistical method as in outcome 11, analysis 1]; Least-squares Mean Difference = -0.6, 95% CI 2-sided [-3.4 to 2.2]

12. Secondary Outcome: Change From Baseline in Global Health Status/QoL Score of the EORTC QLQ-C30
Description: To determine effects on symptoms, functioning, and overall HRQoL of durvalumab in combination with platinum-based chemotherapy (paclitaxel and carboplatin) followed by maintenance durvalumab or durvalumab with olaparib when compared to platinum-based chemotherapy alone in newly diagnosed advanced or recurrent endometrial cancer patients. The global health status/quality of life (QoL) is a score from 0 to 100. Higher scores on the global health status/QoL indicate better health status/function.
Time Frame: as for outcome 11
Population: FAS consisting of all patients randomised as part of global enrolment including patients from China who were randomised before the global recruitment was closed (up to and including 20 Apr 2022). All participants with a baseline and post baseline global health status/QoL available were analysed. This endpoint was not assessed in the China cohort as it was not prespecified in the SAP.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib
Number analyzed (Participants) | 187 | 190 | 199
Score on a scale | -2.8 (0.93) | -2.7 (0.92) | -3.6 (0.88)
Statistical Analysis 1: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab; Test type: Superiority; Mixed model for repeated measures — Descriptive analysis only; [statistical method as in outcome 11, analysis 1]; Least-squares Mean Difference = 0.0, 95% CI 2-sided [-2.5 to 2.6]
Statistical Analysis 2: Comparison: Global Cohort - SoC vs Global Cohort - SoC + Durvalumab + Olaparib; Test type: Superiority; Mixed model for repeated measures — Descriptive analysis only; [statistical method as in outcome 11, analysis 1]; Least-squares Mean Difference = -0.9, 95% CI 2-sided [-3.4 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) with onset date or that worsen on or after first dose of study treatment) up until the initiation of the first subsequent anticancer therapy following discontinuation of study treatment or until the end of safety follow-up period (latest of 30 days following discontinuation of olaparib/placebo or 90 days following discontinuation of durvalumab/placebo), whichever occurs first. DCO: 12 Apr 2023 (08 Jul 2024 for China cohort), up to 50 months
Description: Deaths analysed in FAS; AEs analysed in all randomised patients who received study treatment. MedDRA 25.1 and 27.0 were used to code AEs in the Global and China cohorts, respectively. If the PT is not part of the MedDRA dictionary, the count is presented as zero. Otherwise, zero means that the term is part of the MedDRA version but no events were observed.
  Included in MedDRA 25.1 but not in MedDRA 27.0: Myxoedema coma Included in MedDRA 27.0 but not in MedDRA 25.1: Bile acids increased
Groups:
- China Cohort - SoC: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with durvalumab placebo (IV) Q3W.
  Following completion of chemotherapy treatment, participants without objective disease progression received durvalumab placebo (IV) Q4W and olaparib placebo (tablets) twice bd orally as maintenance treatment until disease progression.
- China Cohort - SoC + Durvalumab: Platinum-based chemotherapy (paclitaxel and carboplatin) Q3W for a maximum of 6 cycles with 1120 mg durvalumab (IV) Q3W.
  Following completion of chemotherapy treatment, participants without objective disease progression received 1500 mg durvalumab (IV) Q4W with olaparib placebo (tablets) bd orally as maintenance treatment until disease progression.
Arm/Group | Global Cohort - SoC | Global Cohort - SoC + Durvalumab | Global Cohort - SoC + Durvalumab + Olaparib | China Cohort - SoC | China Cohort - SoC + Durvalumab | China Cohort - SoC + Durvalumab + Olaparib
All-Cause Mortality (participants affected / at risk) | 82/241 | 65/238 | 52/239 | 12/44 | 11/43 | 14/42
Serious Adverse Events (participants affected / at risk) | 73/236 | 73/235 | 85/238 | 14/44 | 8/41 | 19/41
Other Adverse Events (participants affected / at risk) | 233/236 | 228/235 | 236/238 | 44/44 | 41/41 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort - SoC (N=236) | Global Cohort - SoC + Durvalumab (N=235) | Global Cohort - SoC + Durvalumab + Olaparib (N=238) | China Cohort - SoC (N=44) | China Cohort - SoC + Durvalumab (N=41) | China Cohort - SoC + Durvalumab + Olaparib (N=41)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paracancerous pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
West nile viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 1 (1) | 16 (33) | 1 (6) | 1 (2) | 4 (17)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myxoedema coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary cerebellar degeneration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 4 (4) | 7 (8) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperplasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort - SoC (N=236) | Global Cohort - SoC + Durvalumab (N=235) | Global Cohort - SoC + Durvalumab + Olaparib (N=238) | China Cohort - SoC (N=44) | China Cohort - SoC + Durvalumab (N=41) | China Cohort - SoC + Durvalumab + Olaparib (N=41)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 4 (5) | 11 (12) | 7 (7) | 4 (6) | 4 (6)
Urinary tract infection (Infections and infestations) | 47 (65) | 32 (62) | 46 (67) | 8 (12) | 4 (10) | 5 (8)
Neutropenia (Blood and lymphatic system disorders) | 30 (48) | 34 (61) | 47 (85) | 2 (3) | 3 (4) | 4 (8)
Fall (Injury, poisoning and procedural complications) | 10 (10) | 14 (14) | 15 (19) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 22 (28) | 14 (19) | 12 (17) | 1 (2) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 18 (24) | 30 (37) | 30 (41) | 17 (33) | 16 (28) | 11 (22)
Aspartate aminotransferase increased (Investigations) | 17 (26) | 22 (26) | 20 (25) | 17 (35) | 13 (24) | 14 (26)
Bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 6 (8) | 11 (13) | 8 (9) | 4 (4) | 5 (7) | 5 (6)
Blood bilirubin increased (Investigations) | 4 (7) | 4 (7) | 0 (0) | 5 (8) | 1 (1) | 4 (8)
Blood creatinine increased (Investigations) | 13 (20) | 10 (13) | 24 (42) | 2 (3) | 4 (7) | 10 (21)
Blood lactate dehydrogenase increased (Investigations) | 14 (19) | 9 (15) | 8 (14) | 4 (5) | 5 (8) | 7 (10)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 4 (5) | 3 (4) | 0 (0) | 4 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 4 (5) | 3 (3) | 4 (7) | 2 (5) | 3 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (30) | 30 (49) | 35 (70) | 5 (10) | 3 (6) | 4 (9)
Blood urea increased (Investigations) | 4 (6) | 3 (3) | 3 (4) | 4 (17) | 2 (4) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 12 (14) | 17 (17) | 15 (22) | 8 (12) | 9 (15) | 7 (15)
Hepatic enzyme increased (Investigations) | 5 (12) | 1 (1) | 4 (11) | 3 (10) | 3 (4) | 1 (7)
Lipase increased (Investigations) | 11 (12) | 7 (8) | 5 (6) | 3 (6) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (21) | 11 (17) | 12 (17) | 6 (28) | 7 (24) | 10 (32)
Neutrophil count decreased (Investigations) | 60 (159) | 43 (105) | 50 (145) | 30 (138) | 30 (132) | 29 (149)
Neutrophil count increased (Investigations) | 1 (6) | 2 (2) | 0 (0) | 2 (8) | 3 (4) | 3 (3)
Platelet count decreased (Investigations) | 37 (73) | 36 (61) | 39 (71) | 21 (66) | 13 (24) | 15 (38)
Weight decreased (Investigations) | 23 (28) | 20 (24) | 17 (17) | 6 (8) | 3 (3) | 8 (10)
Weight increased (Investigations) | 7 (7) | 7 (7) | 10 (12) | 5 (5) | 5 (5) | 1 (2)
White blood cell count decreased (Investigations) | 40 (111) | 29 (67) | 38 (112) | 32 (159) | 30 (129) | 31 (161)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 1 (12) | 2 (3) | 3 (4) | 5 (19)
Decreased appetite (Metabolism and nutrition disorders) | 46 (60) | 42 (57) | 55 (83) | 3 (3) | 5 (6) | 10 (18)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (10) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (25) | 8 (12) | 17 (19) | 5 (11) | 7 (9) | 4 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (11) | 5 (6) | 7 (9) | 0 (0) | 3 (5) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (3) | 3 (3) | 3 (3) | 2 (6) | 1 (1) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (13) | 3 (3) | 5 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 0 (0) | 9 (18) | 8 (26) | 4 (17)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (9) | 10 (17) | 4 (8) | 9 (19) | 7 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (6) | 5 (8) | 2 (2) | 3 (3) | 2 (6) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (37) | 26 (42) | 27 (49) | 11 (29) | 7 (12) | 8 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 38 (53) | 38 (49) | 38 (66) | 9 (18) | 5 (8) | 4 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (17) | 8 (11) | 12 (22) | 4 (6) | 2 (2) | 9 (12)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 (89) | 70 (112) | 58 (98) | 5 (5) | 6 (7) | 5 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (33) | 19 (23) | 35 (39) | 3 (3) | 4 (4) | 1 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 16 (19) | 11 (16) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (10) | 8 (9) | 0 (0) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (19) | 15 (17) | 13 (17) | 1 (1) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 44 (73) | 32 (47) | 30 (33) | 1 (1) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 (42) | 31 (44) | 29 (38) | 10 (15) | 6 (13) | 9 (11)
Dizziness (Nervous system disorders) | 30 (38) | 32 (37) | 40 (50) | 3 (3) | 3 (5) | 5 (5)
Dysgeusia (Nervous system disorders) | 26 (27) | 24 (28) | 27 (33) | 1 (1) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 35 (42) | 30 (34) | 39 (49) | 2 (2) | 2 (2) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 12 (19) | 9 (10) | 15 (19) | 16 (24) | 7 (11) | 18 (21)
Anaemia (Blood and lymphatic system disorders) | 121 (160) | 111 (168) | 141 (242) | 36 (101) | 28 (70) | 34 (88)
Neuropathy peripheral (Nervous system disorders) | 66 (83) | 61 (69) | 60 (74) | 2 (2) | 4 (5) | 2 (2)
Paraesthesia (Nervous system disorders) | 10 (11) | 13 (14) | 6 (9) | 2 (2) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 66 (74) | 60 (69) | 60 (66) | 2 (2) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 33 (35) | 24 (28) | 29 (31) | 6 (8) | 7 (9) | 5 (6)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (5)
Dysuria (Renal and urinary disorders) | 12 (16) | 10 (12) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 11 (11) | 4 (4) | 7 (8) | 1 (1) | 3 (3) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 15 (15) | 3 (3) | 9 (11) | 1 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 4 (7) | 4 (5) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 13 (15) | 11 (12) | 9 (9) | 1 (1) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 35 (38) | 32 (40) | 2 (2) | 9 (11) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 27 (34) | 29 (36) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 118 (118) | 118 (122) | 121 (124) | 29 (29) | 20 (20) | 26 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (41) | 36 (42) | 37 (58) | 6 (12) | 2 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 27 (32) | 41 (59) | 28 (38) | 6 (6) | 11 (33) | 7 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 13 (16) | 15 (23) | 1 (2) | 3 (5) | 0 (0)
Hypertension (Vascular disorders) | 13 (18) | 10 (10) | 13 (27) | 4 (8) | 1 (1) | 3 (17)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 15 (16) | 13 (15) | 1 (1) | 4 (4) | 6 (7)
Hypothyroidism (Endocrine disorders) | 8 (9) | 37 (44) | 33 (42) | 4 (4) | 10 (12) | 5 (10)
Vision blurred (Eye disorders) | 10 (10) | 12 (15) | 9 (9) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 11 (12) | 10 (17) | 13 (15) | 3 (3) | 3 (6) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 38 (39) | 38 (49) | 40 (53) | 3 (4) | 5 (14) | 4 (8)
Abdominal pain lower (Gastrointestinal disorders) | 13 (13) | 8 (9) | 6 (7) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (12) | 16 (17) | 14 (16) | 4 (5) | 4 (7) | 1 (2)
Constipation (Gastrointestinal disorders) | 80 (102) | 63 (80) | 78 (105) | 10 (10) | 5 (9) | 11 (18)
Diarrhoea (Gastrointestinal disorders) | 64 (101) | 74 (115) | 67 (114) | 10 (13) | 2 (2) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 5 (5) | 9 (14) | 0 (0) | 0 (0) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 18 (21) | 12 (13) | 22 (28) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 105 (182) | 95 (157) | 129 (237) | 18 (30) | 11 (30) | 18 (60)
Stomatitis (Gastrointestinal disorders) | 18 (24) | 19 (20) | 25 (31) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 7 (8) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 42 (72) | 46 (73) | 61 (93) | 11 (15) | 11 (25) | 18 (37)
Asthenia (General disorders) | 23 (34) | 22 (31) | 44 (72) | 0 (0) | 1 (1) | 3 (8)
Chest discomfort (General disorders) | 4 (5) | 4 (4) | 5 (7) | 2 (3) | 3 (3) | 1 (2)
Fatigue (General disorders) | 87 (127) | 82 (101) | 93 (143) | 4 (4) | 2 (2) | 6 (8)
Influenza like illness (General disorders) | 8 (9) | 10 (14) | 9 (9) | 2 (2) | 6 (6) | 2 (3)
Malaise (General disorders) | 16 (21) | 14 (31) | 12 (18) | 3 (3) | 5 (5) | 9 (13)
Oedema peripheral (General disorders) | 21 (23) | 29 (35) | 30 (37) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 9 (14) | 6 (6) | 10 (14) | 3 (6) | 3 (3) | 5 (8)
Peripheral swelling (General disorders) | 6 (6) | 8 (8) | 10 (12) | 1 (2) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 18 (20) | 20 (27) | 23 (30) | 2 (2) | 4 (6) | 7 (10)
Leukocytosis (Blood and lymphatic system disorders) | 3 (6) | 4 (4) | 1 (2) | 2 (6) | 3 (3) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 9 (14) | 12 (25) | 15 (37) | 3 (6) | 6 (25) | 7 (22)
Covid-19 (Infections and infestations) | 29 (29) | 35 (36) | 44 (46) | 6 (8) | 8 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT04269200/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04269200/SAP_001.pdf